CLINICAL TRIAL: NCT03043664
Title: Phase Ib/II Study of Pembrolizumab With Lanreotide Depot for Gastroenteropancreatic Neuroendocrine Tumors
Brief Title: Study of Pembrolizumab With Lanreotide Depot for Gastroenteropancreatic Neuroendocrine Tumors
Acronym: PLANET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00074917
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors
Keywords: GEP-NET; pembrolizumab; lanreotide; PD-1; Keytruda; Somatuline Depot; PD-L1; anti-PD-1
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — lanreotide; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Keytruda (pembrolizumab) 200 mg intravenous (IV) infusion every 3 weeks and Somatuline Depot (lanreotide) 90 mg subcutaneous (SQ) injection every 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Keytruda (pembrolizumab) 200 mg intravenous (IV) infusion every 3 weeks and Somatuline Depot (lanreotide) 90 mg subcutaneous (SQ) injection every 3 weeks.
  Interventions: Drug: Lanreotide; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lanreotide — Somatuline depot (lanreotide) 90 mg SQ every 3 weeks
  Other Names: Somatuline Depot
Drug: Pembrolizumab — Keytruda (pembrolizumab) 200 mg IV every 3 weeks
  Other Names: Keytruda

SUMMARY:
This study is for patients with non-resectable, recurrent, or metastatic well or moderately differentiated gastroenteropancreatic neuroendocrine tumors (GEP-NETs).

The study will be conducted in two stages: 1) Safety Run-In and 2) Expanded Cohort.

1. Safety run-in: The first stage will include a safety run-in of 6 patients treated with pembrolizumab 200 mg intravenous (IV) every 3 weeks and lanreotide depot 90mg subcutaneous (SQ) every 3 weeks. Up to 6 patients at the Duke Cancer Institute will be accrued at the starting dose level. If one or less subject meets treatment-related discontinuation criteria (as specified in the protocol) during Cycle 1, then the study will proceed to the second stage, Expanded Cohort.
2. Expanded Cohort: Patients will be treated with pembrolizumab 200mg IV every 3 weeks and lanreotide depot 90mg SQ every 3 weeks as determined by the Safety Run-In Cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the trial.
2. At least 18 years of age on day of signing informed consent.
3. Non-resectable, recurrent, or metastatic well- or moderately-differentiated gastroenteropancreatic neuroendocrine tumor (GEP-NETs) with disease progression within the last 12 months. (Patients who have received prior local therapy, including but not limited to embolization, chemoembolization, radiofrequency ablation, radiation therapy, are eligible provided that measurable disease falls outside the treatment field or within the field but has shown an increase of > 20% in the size. Prior local therapy must be completed at least 4 weeks prior to the baseline scan.)
4. Prior somatostatin analogue therapy. (Patients should receive the first dose of study drug no sooner than 4 weeks from the last dose of somatostatin analogue.)
5. At least one measurable lesion based on RECIST version 1.1.
6. Agrees to provide available archived tumor tissue specimen. (Patients who do not have available archived tumor must agree to have core or excisional biopsy of a tumor lesion obtained up to 42 days prior to the first dose of study drug, if safely accessible. If archived tissue is not available and the tumor is not amenable to safe biopsy, subject is still eligible to participate.)
7. ECOG performance status of 0 or 1.
8. Adequate organ function defined as:

   * Absolute neutrophil count (ANC) ≥ 1,500 /mcL
   * Platelets ≥ 100,000 /mcL
   * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
   * Serum creatinine OR calculated creatinine clearance (CrCL) per institutional standard (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 X upper limit of normal (ULN) OR ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
   * Serum total bilirubin ≤ 1.5 X ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
   * Albumin ≥ 2.5 mg/dL
9. Negative serum pregnancy test within ≤ 7 days prior to the first dose of study drug, for women of childbearing potential only.
10. Female subjects agree to use two birth control methods, be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study drug.
11. Male subjects agree to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Tumor mitotic rate >20/10 hpf and/or Ki67 index >20% (if available).
2. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
3. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
4. Known history of active TB (Bacillus Tuberculosis).
5. Hypersensitivity to pembrolizumab or lanreotide or any of their excipients.
6. Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to the first dose of study drug or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
7. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of study drug or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Patients with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
8. Prior major surgery within 2 weeks prior to the first dose of study drug or who has not recovered adequately from the toxicity and/or complications from the intervention.
9. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
10. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to the first dose of study drug. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
11. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Known history of, or any evidence of active, non-infectious pneumonitis.
13. Active infection requiring systemic therapy.
14. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating physician.
15. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of study drug.
17. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
18. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
20. Live vaccine within 30 days of planned start of study drug regimen. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
21. History of intolerance to somatostatin analogues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morse, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Lexington Medical Center, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Duke University Medical Center from 5/15/2017 to 2/13/2020.
Groups:
- Somatuline Depot and Keytruda: Keytruda (pembrolizumab) 200 mg intravenous (IV) infusion every 3 weeks and Somatuline Depot (lanreotide) 90 mg subcutaneous (SQ) injection every 3 weeks.
Period: Overall Study
Arm/Group | Somatuline Depot and Keytruda
Started | 22
Completed | 21
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Somatuline Depot and Keytruda
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 9
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR is calculated as the number of people with a complete response (CR) or partial response (PR), divided by the total number of people treated. Complete response is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. A lower limit of the true ORR will be estimated by the 90% exact lower confidence bound (LCB) for the binomial proportion. A 90% LCB of < 0.1 will be considered not to be of clinical value. If the 90% LCB is ≥ 0.1, the regimen will be considered efficacious.
Time Frame: Approximately every 12 weeks until study completion (up to 2 years)
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Somatuline Depot and Keytruda
Number analyzed (Participants) | 22
proportion of participants | 0.045 [0 to 0.12]

2. Secondary Outcome: Number of Participants Experiencing Treatment-related AEs Leading to Drug Discontinuations During the First 12 Weeks of Treatment
Description: Adverse events were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: First 12 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Somatuline Depot and Keytruda
Number analyzed (Participants) | 22
Participants | 0

3. Secondary Outcome: Months of Progression-free Survival (PFS)
Description: Months from treatment start date until the date of first documented radiographic progression or date of death from any cause (whichever is first); assessed up to 48 weeks after the last subject has finished study drug regimen. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Somatuline Depot and Keytruda
Number analyzed (Participants) | 22
months | 5.04 [2.7 to 11.3]

4. Secondary Outcome: Months of Overall Survival (OS)
Description: Months from treatment start date until the date of death from any cause; assessed up to 48 weeks after the last subject has finished the study drug regimen
Time Frame: Up to 59 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Somatuline Depot and Keytruda
Number analyzed (Participants) | 22
months | 28.6 [21.0 to NA] — There is not a sufficient number of events after the median time point to estimate the upper confidence limit. Most patients past the median are censored.

5. Secondary Outcome: ORR as Measured by Immune-related Response Criteria (irRC)
Description: Treatment response as assessed by irRC instead of RECIST v1.1. ORR is calculated as the number of people with a complete response (CR) or partial response (PR), divided by the total number of people treated. Complete response is defined as complete disappearance of all lesions (whether measurable or not, and no new lesions), confirmed by a repeat, consecutive assessment no less than 4 weeks from the date first documented. Partial response is defined as a decrease in tumor burden ≥ 50% relative to baseline, confirmed by a consecutive assessment at least 4 weeks after first documentation. A lower limit of the true ORR will be estimated by the 90% exact lower confidence bound (LCB) for the binomial proportion.
Time Frame: Approximately every 12 weeks until study completion (up to 2 years)
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Somatuline Depot and Keytruda
Number analyzed (Participants) | 22
proportion of participants | 0.045 [0 to 0.12]

ADVERSE EVENTS:
Time Frame: Up to 25 months for adverse events; up to 59 months for all-cause mortality
Arm/Group | Somatuline Depot and Keytruda
All-Cause Mortality (participants affected / at risk) | 15/22
Serious Adverse Events (participants affected / at risk) | 6/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatuline Depot and Keytruda (N=22)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4)
Colitis (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (2)
Infections and infestations - Other, Specify, Salmonella (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatuline Depot and Keytruda (N=22)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 5 (5)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Ascites (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 12 (12)
Injection site reaction (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, Specify, Non Fasting Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Specify, Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03043664/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT03043664/ICF_001.pdf